CLINICAL TRIAL: NCT03335358
Title: Pilot Testing a Positive Psychology-based Intervention for Couples Coping With Stroke: Promoting Resilience After Stroke in Dyads (RESToreD)
Brief Title: Testing a Positive Psychology-based Intervention for Couples Coping With Stroke
Acronym: RESToreD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Alexandra Terrill, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1R03HD091432-01 (NIH)
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Stroke; Depression; Depressive Symptoms; Post-stroke Depression
Keywords: couples; positive psychology; behavioral intervention; stroke; depression; wellbeing; caregiver
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Intervention Model Description: Waitlist control design; participants are assigned to receive intervention or be waitlisted for 4-6 weeks and then receive intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Intervention (Experimental): Participants complete baseline assessments and receive a 20min training on the positive psychology activities. They are instructed to engage in at least 2 positive psychology activities alone and at least 2 as a couple each week for 8 weeks. Self-administered activities include expressing gratitude, practicing acts of kindness, focusing on the positive, fostering relationships, working toward a goal, spirituality, savoring. Post-intervention and 3-month follow-up assessments are completed.
  Interventions: Behavioral: Dyadic (couples-based) positive psychology intervention
- Waitlist control (Other): Participants complete a baseline assessment and are waitlisted for 4-6 weeks. They then complete another assessment, receive the 20min training on activities, and then complete the 8-week self-administered intervention (same as the experimental arm). Post-intervention and 3-month follow up assessments are also completed.
  Interventions: Behavioral: Dyadic (couples-based) positive psychology intervention

INTERVENTIONS:
Behavioral: Dyadic (couples-based) positive psychology intervention — Self-administered behavioral intervention in which participants complete at least 2 activities alone and 2 together each week for 8 weeks. Positive psychology activities include expressing gratitude, practicing acts of kindness, fostering relationships, working toward a goal, focusing on the positive, spirituality, and savoring.

SUMMARY:
This study aims to pilot test an 8-week, self-administered dyadic (couples-based) positive psychology intervention for couples coping with stroke using a randomized, waitlist control design. Mood and well-being will be assessed pre- and post-intervention, and at 3-month follow-up. It is expected that both partners will demonstrate improvement in mood and well-being.

DETAILED DESCRIPTION:
Stroke survivors and spousal caregivers face significant challenges, yet interventions to support couples after stroke are largely lacking. Depressive symptoms post-stroke occur in 30-50% of survivors and partner caregivers, and have significant consequences on function and quality of life. Further, mood and psychosocial well-being are reciprocal in couples, meaning if one partner is depressed, the other is more likely to be depressed. Sustaining well-being in both partners is important for continued engagement in rehabilitation and re-integration into the community, yet existing interventions are aimed at the individual rather than the couple. This study will address this gap by testing an innovative dyadic (couples-based) intervention using a new approach based on positive psychology that focuses on the strengths in the relationship in order to foster resilience in the couple. Using a randomized waitlist control design, this pilot study aims to determine whether an 8-week dyadic positive psychology-based intervention (PPI) can improve mood and subjective well-being as assessed by established outcome measures in 24 couples coping with stroke. The intervention consists of self-administered PPI activities, such as expressing gratitude and practicing acts of kindness, which participants complete individually and as a couple. Two potential pathways will be explored for the PPI: (a) enhanced quality of interactions as couples deal with daily life demands and (b) improvements in mood that are "contagious" among couples. If found effective, couples with greater well-being may be better emotionally equipped to cope with the sequelae of stroke by reducing stress and depressive symptoms, and increasing participation in meaningful activities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Couples consist of one partner who had an ischemic or hemorrhagic stroke >3 months ago and a cohabiting partner (> 1 year) who self-identifies as the caregiver and is willing to enroll in the study;
* Either one or both partner(s) report depressive symptoms as assessed by the PROMIS-D (no formal diagnosis is required).

Exclusion Criteria:

* the caregiver has had a stroke or other major neurological condition;
* either partner is unable to understand the printed English instructions;
* either partner scores <19 (the established cut-off for mild cognitive impairment) on the Montreal Cognitive Assessment (MoCA), a validated screening instrument for cognitive performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
PROMIS Depression-SF | Change from baseline to 8 weeks (post-intervention)
  An 8-item measure of depressive symptoms in which participants rate how they have felt over the past 7 days (e.g., "I felt worthless," "I felt unhappy") on a 5-point Likert scale from "never" to "always"). Higher scores are worse.
NeuroQOL Positive Affect and Wellbeing-SF | Change from baseline to 8 weeks (post-intervention)
  A 9-item measure of wellbeing in which participants rate how they have felt "lately" (e.g., "my life had purpose," "I felt hopeful") on a 5-point Likert scale from "never" to "always". Higher scores are better
NeuroQOL Positive Affect and Wellbeing-SF | Change from 8 weeks to 20 weeks (3-months post-intervention)
  A 9-item measure of wellbeing in which participants rate how they have felt "lately" (e.g., "my life had purpose," "I felt hopeful") on a 5-point Likert scale from "never" to "always". Higher scores are better
PROMIS Depression-SF | Change from 8 weeks to 20 weeks (3-months post-intervention)
  An 8-item measure of depressive symptoms in which participants rate how they have felt over the past 7 days (e.g., "I felt worthless," "I felt unhappy") on a 5-point Likert scale from "never" to "always"). Higher scores are worse.

SECONDARY OUTCOMES:
Stroke Impact Scale | Change from baseline to 8 weeks (post-intervention)
  A 60-item stroke-specific quality of life measure in which participants rate how stroke has impacted them across 8 domains (e.g., strength of affected arm, communication, activities of daily living) on a 5-point Likert scale ("not difficult" to "cannot do at all"). Higher scores are better (indicate better quality of life)
Stroke Impact Scale | Change from 8 weeks (post-intervention) to 20 weeks (3-months post-intervention)
  A 60-item stroke-specific quality of life measure in which participants rate how stroke has impacted them across 8 domains (e.g., strength of affected arm, communication, activities of daily living) on a 5-point Likert scale ("not difficult" to "cannot do at all"). Higher scores are better (indicate better quality of life)
Positive Affect and Negative Affect Schedule (PANAS) | Change from baseline to 8 weeks (post-intervention)
  A measure of positive affect and negative affect; participants rate a list of 20 adjectives that describes them (e.g., "afraid" or "excited") on a 5-point Likert scale from "Not at all" to "Extremely". Scores are summed for two subscales (positive affect, negative affect), and higher scores indicate having more of either positive or negative affect
Positive Affect and Negative Affect Schedule (PANAS) | Change from 8 weeks (post-intervention) to 20 weeks (3-months post-intervention)
  A measure of positive affect and negative affect; participants rate a list of 20 adjectives that describes them (e.g., "afraid" or "excited") on a 5-point Likert scale from "Not at all" to "Extremely". Scores are summed for two subscales (positive affect, negative affect), and higher scores indicate having more of either positive or negative affect

OTHER OUTCOMES:
Caregiver Strain Index | Change from baseline to 8 weeks (post-intervention)
  A 13-item measure of caregiver strain, in which participants respond yes (1 point) or no (0 points) to items including "sleep is disturbed," and "it is inconvenient"; higher scores mean more strain
Caregiver Strain Index | Change from 8 weeks (post-intervention) to 20 weeks (3-months post-intervention)
  A 13-item measure of caregiver strain, in which participants respond yes (1 point) or no (0 points) to items including "sleep is disturbed," and "it is inconvenient"; higher scores mean more strain
Dyadic Coping Inventory | Change from baseline to 8 weeks (post-intervention)
  A 39-item measure of coping for couples in which participants indicate how they (as a couple) cope with stress on a 5-item Likert scale from "very rarely" to "very often". Higher scores indicate better/more adaptive coping
Dyadic Coping Inventory | Change from 8 weeks (post-intervention) to 20 weeks (3-months post-intervention)
  A 39-item measure of coping for couples in which participants indicate how they (as a couple) cope with stress on a 5-item Likert scale from "very rarely" to "very often". Higher scores indicate better/more adaptive coping

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Terrill, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all outcome measures will be made available. The data will be made available within 1 year of study completion. Access requests will be reviewed, and a data access agreement is required.

REFERENCES:
- [Result] Terrill AL, Reblin M, MacKenzie JJ, Cardell B, Einerson J, Berg CA, Majersik JJ, Richards L. Development of a novel positive psychology-based intervention for couples post-stroke. Rehabil Psychol. 2018 Feb;63(1):43-54. doi: 10.1037/rep0000181. PMID 29553781
- [Derived] Terrill AL, Reblin M, MacKenzie JJ, Baucom BRW, Einerson J, Cardell B, Richards L, Majersik JJ. Promoting Resilience After Stroke in Dyads (ReStoreD): A Supplemental Analysis. Arch Phys Med Rehabil. 2023 Oct;104(10):1580-1587. doi: 10.1016/j.apmr.2023.03.024. Epub 2023 Apr 17. PMID 37075965
- [Derived] Einerson J, Lundstrom LK, Allen BK, Sefandonakis A, Terrill AL. Learning to flourish in a new reality: a thematic analysis of couples' experience of participation in a positive psychology intervention post-stroke. Disabil Rehabil. 2023 Aug;45(16):2612-2619. doi: 10.1080/09638288.2022.2102256. Epub 2022 Aug 1. PMID 35914538
- [Derived] Niermeyer M, Einerson J, Terrill AL. Perceptions of function and recovery among persons with stroke and care partners. Rehabil Psychol. 2022 May;67(2):215-225. doi: 10.1037/rep0000441. Epub 2022 Apr 4. PMID 35377699
- [Derived] Terrill AL, Reblin M, MacKenzie JJ, Baucom BRW, Einerson J, Cardell B, Richards LG, Majersik JJ. Intimate Relationships and Stroke: Piloting a Dyadic Intervention to Improve Depression. Int J Environ Res Public Health. 2022 Feb 5;19(3):1804. doi: 10.3390/ijerph19031804. PMID 35162827
- [Derived] Anderson MA, Buffo C, Ketcher D, Nguyen H, MacKenzie JJ, Reblin M, Terrill AL. Applying the RISE Model of Resilience in Partners Post-Stroke: A Qualitative Analysis. Ann Behav Med. 2022 Mar 1;56(3):270-281. doi: 10.1093/abm/kaab053. PMID 34228090

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03335358/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03335358/ICF_001.pdf